CLINICAL TRIAL: NCT06234449
Title: The Impact of Long-term Pessary Use on Pelvic Organ Prolapse oìduring Covid-19 Pandemic in Patients Attending Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Stefano Salvatore, Professor, IRCCS San Raffaele
Other Study IDs: POP-ES
Record Dates: First submitted 2024-01-25; First posted 2024-01-31 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Pelvic Organ Prolapse; Vaginal Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Vaginal pessary before surgery for pelvic organ prolapse — use of vaginal pessary for patients waiting for gynecological surgery for stage III and IV pelvic organ prolapse

SUMMARY:
Patients aged 45 to 80 years with a clinical diagnosis of stage III and IV genital prolapse involving the anterior and/or middle compartments and candidates for surgery will be considered. These will be evaluated to observe whether there is improvement in clinical prolapse with the use of the vaginal pessary during the waiting period for surgery

ELIGIBILITY:
Inclusion Criteria:

* Pelvic organ prolapse with POP-Q stage >/= 3 in anterior and/or central compartments
* Women between 45 and 80 years old

Exclusion Criteria:

* Women who refuse to participate in the study
* Patients without baseline POPQ examination documented or with a pessary previously positioned
* Previous pelvic surgeries
* Women with any contraindication for surgery or preference for conservative treatment only (pelvic muscle exercise, vaginal pessary)
* Women who are not successfully fitted with pessaries
* Current genital ulcers/infections
* Active or chronic pelvic infection
* Women who are mentally incapable of completing the questionnaires.

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with symptomatic and documented POP (stages III and IV) through POPQ examination who opted for reconstructive surgery and managed with pessary until surgery will be included in the cohort.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
evaluate a change in POPQ points on examination at the time of surgery from baseline evaluation. | At the time of surgery procedure, after at least 6 months after pessary placement
  Primary endopoint is the evaluation of the percentage of women who experience a change in any POPQ point on examination at the time of surgery from baseline evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided